CLINICAL TRIAL: NCT02719327
Title: Impact of Icosapent Ethyl on Alzheimers Disease Biomarkers in Preclinical Adults
Brief Title: Brain Amyloid and Vascular Effects of Eicosapentaenoic Acid
Acronym: BRAVE-EPA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLNA-001-15S; CX001261 (Other Grant/Funding Number: VA Merit)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Cerebrospinal fluid; brain blood flow; cognition; icosapent ethyl; Vascepa; omega-3 fatty acids; eicosapentaenoic acid
MeSH Terms: conditions — Alzheimer Disease | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of icosapent ethyl 4 g daily vs matching placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- icosapent ethyl (IPE) (Experimental): Participants will be randomized in a 1:1 ratio to receive icosapent ethyl 4 g daily vs. matching gel cap placebo
  Interventions: Drug: icosapent ethyl (IPE)
- placebo (Placebo Comparator): Participants will be randomized in a 1:1 ratio to receive icosapent ethyl 4 g daily vs. matching gel cap placebo
  Interventions: Other: gel cap placebo

INTERVENTIONS:
Drug: icosapent ethyl (IPE) — Participants will be randomized in a 1:1 ratio to receive icosapent ethyl 4 g daily vs. matching gel cap placebo
  Other Names: Vascepa
  Arms: icosapent ethyl (IPE)
Other: gel cap placebo — Participants will be randomized in a 1:1 ratio to receive icosapent ethyl 4 g daily vs. matching gel cap placebo
  Other Names: Placebo
  Arms: placebo

SUMMARY:
The number of Americans diagnosed with Alzheimer's disease (AD) is expected to triple by 2050. Compared to the general population, Veterans have a greater risk of AD, likely in part due to their increased incidence of traumatic brain injury, post-traumatic stress disorder, depression, and other vascular-related health issues. Based on available data, 423,000 new cases of AD are anticipated in Veterans by 2020. Thus, the discovery of effective therapies to prevent or delay the onset of AD in Veterans is critical. The goal of this study is to evaluate the efficacy of a purified form of the omega-3 fatty acid eicosapentaenoic acid (EPA) called icosapent ethyl (IPE), on improving brain blood flow, spinal fluid markers of AD pathology, and cognitive performance in middle-aged, cognitively-healthy Veterans with increased risk of AD. If IPE delays the onset of AD by even 5 years, the incidence of AD would be reduced by 50% in this population and could have a profound effect on Veteran quality of life and healthcare costs.

DETAILED DESCRIPTION:
The proposed study is a proof-of-concept, randomized, placebo-controlled, double-blind, parallel-group clinical trial assessing the efficacy of 18 months of icosapent ethyl (IPE) therapy on magnetic resonance imaging (MRI), cerebrospinal fluid (CSF), and cognitive biomarkers for AD in 150 cognitively-healthy Veterans ages 50-75 years. The overarching goal of this trial is to assess whether icosapent ethyl beneficially affects intermediate physiological measures associated with onset of AD in order to evaluate whether larger, multi-site, longer-duration Alzheimer's prevention trials are warranted to assess more definitive clinical outcomes. The proposed study aims to: 1) investigate the effects of 18 months of IPE vs. placebo on regional cerebral blood flow as measured by arterial spin-labeling MRI; 2) determine the impact of 18 months of IPE vs. placebo on CSF biomarkers of AD pathology; and 3) evaluate the effects of 18 months of IPE vs. placebo on cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* United States Veteran eligible for VA care
* Age 50-75 years, inclusive
* Cognitively healthy

Exclusion Criteria:

* Dementia or mild cognitive impairment on screening evaluation
* Current use of fish oil supplements (requires 3 month wash-out period)
* Active liver disease with AST or ALT greater than twice the upper limit of normal
* Elevated creatine kinase greater than twice the upper limit of normal
* Prior adverse reaction to statins or fish oil
* Pregnant, nursing, or pregnancy planned
* Use of medications that interact with icosapent ethyl
* Current use of anticoagulants
* Known hypersensitivity to fish and/or shellfish
* Current use of other investigational drug
* History of significant atherosclerotic cardiovascular disease or diabetes mellitus
* Low-density lipoprotein (LDL) cholesterol > or =190 mg/dL or <80 mg/dL
* Triglycerides > or = 500 mg/dL
* Creatinine >1.8 mg/dL
* Previous lumbar surgery with contraindication to lumbar puncture
* Claustrophobia requiring sedation for MRI
* Pacemaker or other contraindication for MRI
* Consumption of >200 mg per day omega-3 fatty acids in diet

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M. Carlsson, MD MS, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Icosapent Ethyl (IPE) | Placebo
Started | 63 | 68
Completed | 52 | 60
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Icosapent Ethyl (IPE) | Placebo | Total
Number analyzed (Participants) | 63 | 68 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.06) | 65.4 (7.00) | 65.5 (7.00)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 52 | 60 | 112
  Unknown | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 61 | 65 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  GED or ABE certificate | 1 | 2 | 3
  High school diploma | 8 | 10 | 18
  Trade or technical school graduate | 8 | 3 | 11
  Some college but not a 2- or 4-year degree | 12 | 15 | 27
  2-year college degree (AA or equivalent) | 14 | 8 | 22
  4-year college degree (Bachelor's) | 11 | 17 | 28
  Master's degree | 8 | 12 | 20
  Did not graduate from high school | 0 | 1 | 1
  Unknown | 1 | 0 | 1
APOE risk allele [Count of Participants; unit: Participants] — Apolipoprotein e4 risk allele carriership.
  Participants
    Carrier | 11 | 19 | 30
    Non-Carrier | 52 | 49 | 101
Parental history of Alzheimer's disease [Count of Participants; unit: Participants]
  Yes | 29 | 32 | 61
  No | 33 | 36 | 69
  Unknown | 1 | 0 | 1
Systolic blood pressure [Mean (Standard Deviation); unit: mm/Hg] | 136.2 (16.4) | 136.1 (16.5) | 136.1 (16.4)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 173.2 (41.4) | 168.3 (45.2) | 170.6 (43.3)

OUTCOME MEASURES:

1. Primary Outcome: Regional Cerebral Blood Flow Using Arterial Spin-labeling MRI
Description: For the primary outcome we chose an anatomical region, posterior cingulate gyrus, that aligned with statistical region of interest sensitive to changes in cerebral blood flow in cognitively-unimpaired adults at risk for Alzheimer's disease. Brain blood flow was averaged across the right and left posterior cingulate gyrus.
Time Frame: 18 month study visit
Population: Analysis sample is intent-to-treat (ITT), ASL values were imputed from baseline values for 23 participants (n=14 IPE and n=9 placebo); 17 participants lacked baseline ASL values (n=9 IPE, n=8 placebo) and could not be included in analyses.
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | Icosapent Ethyl (IPE) | Placebo
Number analyzed (Participants) | 54 | 60
mL/g/min | 55.7 (14.6) | 54.5 (14.1)
Statistical Analysis 1: Comparison: Icosapent Ethyl (IPE) vs Placebo; The proposed study aims to investigate the effects of 18 months of IPE vs. placebo on regional cerebral blood flow in the bilateral posterior cingulate gyrus as measured by arterial spin-labeling MRI . IPE was hypothesized to improve regional cerebral blood flow over placebo after 18 months; Test type: Superiority; p = 0.17, Regression, Linear — ASL values at 18 months were regressed on treatment group (IPE vs placebo) statistically controlling for age at baseline visit and ASL measured at baseline visit; Slope = -2.18, 95% CI 2-sided [-5.36 to 0.99]

2. Secondary Outcome: Cerebrospinal Fluid (CSF) Biomarkers of Alzheimer's Disease
Description: CSF beta-amyloid-42, total tau, and phosphorylated tau-181 (Roche Cobas Elecsys e611). Lower CSF beta-amyloid-42 and higher phosphorylated tau-181 or total tau are associated with risk for Alzheimer's disease.
Time Frame: 18 month study visit
Population: Analysis is based on an intent-to-treat, n=19 participants dropped out prior to receiving an 18 month lumbar puncture (n=11 IPE, n=8 placebo); 26 participants opted out of the lumbar puncture procedure (n=11 IPE, n=15 placebo)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Icosapent Ethyl (IPE) | Placebo
Number analyzed (Participants) | 41 | 45
pg/mL
  beta-amyloid(1-42) | 1281.7 (558.5) | 1244.6 (607.7)
  phosphorylated tau(181) | 20.2 (8.13) | 18.8 (5.56)
  Total tau | 218.2 (83.6) | 208.0 (63.7)
Statistical Analysis 1: Comparison: Icosapent Ethyl (IPE) vs Placebo; Beta-amyloid(1-42) concentration in CSF was log-transformed prior to analysis to approximate a normal distribution; Test type: Superiority; p = .12, Regression, Linear; 18 month Beta-amyloid(1-42) was regressed on group (IPE vs placebo) and covariates age at baseline visit and Beta-amyloid(1-42) at baseline visit; Slope = 0.11, 95% CI 2-sided [-0.04 to 0.25] — Placebo group is the reference group
Statistical Analysis 2: Comparison: Icosapent Ethyl (IPE) vs Placebo; Phosphorylated tau (pTau181) measured in CSF was log-transformed prior to analysis to approximate a normal distribution; Test type: Superiority; p = 0.05, Regression, Linear; log-transformed 18 month pTau181 was regressed on group (IPE vs placebo) and covariates age at baseline and log-transformed ptau181at baseline visit; Slope = 0.045, 95% CI 2-sided [0.004 to 0.061] — Placebo group is the reference group
Statistical Analysis 3: Comparison: Icosapent Ethyl (IPE) vs Placebo; Total tau was log-transformed prior to analysis to better approximate a normal distribution; Test type: Superiority; p = .07, Regression, Linear — 18 months total Tau was regressed on Group (IPE vs placebo) and covariates age at baseline and total Tau at baseline; Slope = 0.046, 95% CI 2-sided [-0.0008 to 0.106] — Placebo group was the reference group

3. Secondary Outcome: Cognitive Performance
Description: Alzheimer's Disease Cooperative Study Preclinical Alzheimer's Cognitive Composite (ADCS-PACC). Composite scores at each time point are standardize to baseline values such that at baseline the mean=0 and the standard deviation = 1. Standardized scores range from -3.15 to 3.09. Higher scores indicate better cognition.
Time Frame: 18 month study visit
Population: Analyses were conducted on an intent-to-treat basis. 19 participants dropped out prior to month 18 study visit (n=11 IPE, n=8)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Icosapent Ethyl (IPE) | Placebo
Number analyzed (Participants) | 52 | 60
Z-score | 0.455 (1.22) | 0.611 (1.10)
Statistical Analysis 1: Comparison: Icosapent Ethyl (IPE) vs Placebo; Four cognitive tests were standardized (baseline mean and standard deviation) prior to averaging to create the ADCS Preclinical Alzheimer Cognitive Composite (ADCS-PACC) score. The final composite score was standardized again using baseline mean and standard deviation (range -3.15 to 3.10). Higher scores indicate better cognitive performance. A linear mixed effects model was used to determine if change in ADCS-PACC composite scores was modified by treatment group; Test type: Superiority; p = .48, Linear Mixed Effects model; Covariates included education level, gender, and age at baseline visit; Slope = 0.006, 95% CI 2-sided [-0.009 to 0.023] — Placebo group was the reference group

ADVERSE EVENTS:
Time Frame: 18 months
Description: Participants were assessed for adverse events at months 1, 3, 6, 9, 12, 15, and 18.
Arm/Group | Icosapent Ethyl (IPE) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 1/68
Serious Adverse Events (participants affected / at risk) | 9/63 | 7/68
Other Adverse Events (participants affected / at risk) | 13/63 | 19/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icosapent Ethyl (IPE) (N=63) | Placebo (N=68)
Mortatilty (General disorders) | 0 (0) | 1 (1) — Participant passed away after falling down a staircase.
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant was hospitalized after COPD attack
Chest pain or tightness (Cardiac disorders) | 1 (1) | 0 (0) — Participant was admitted to hospital after presenting chest tightness
Laparoscopic prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — Participant had planned surgery for prostate cancer.
Surgery (Cardiac disorders) | 1 (1) | 0 (0) — Participant underwent bypass surgery
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Participant admitted after presenting to hospital with heart palpitations.
Aortic aneurysm (Cardiac disorders) | 1 (1) | 0 (0) — Participant admitted to hospital after an aortic aneurysm
non-ST elevated myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Participant hospitalized after a NSTEMI.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant hospitalized after developing spontaneous pneumothorax.
Throat infection (General disorders) | 0 (0) | 1 (1) — Participant hospitalized after presenting with neck pain and inability to swallow.
Dehydration (General disorders) | 1 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Participant presented to the hospital after a fall.
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant was admitted to hospital after developing a UTI.
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Participant hospitalized after presenting with high blood pressure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icosapent Ethyl (IPE) (N=63) | Placebo (N=68)
Headache (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) — Participant reported headache following an LP
Accident (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) — Participant suffered an accidental injury, resolved.
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Synovial cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Participant had a synovial cyst removed from spine (L4/L5).
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported sweating and itching after starting study drug.
Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Resolved.
Distended bladder (Renal and urinary disorders) | 1 (1) | 0 (0) — Resolved.
Hematoma (Renal and urinary disorders) | 0 (0) | 1 (1) — Hematoma following orchiectomy was resolved.
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant fell after feeling light-headed.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitus, eye (Infections and infestations) | 1 (1) | 0 (0)
COVID19 (Infections and infestations) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cancer (Reproductive system and breast disorders) | 1 (1) | 2 (2) — Prostate cancer
Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Positive Colorectal screening
Sinus infection (Infections and infestations) | 1 (1) | 0 (0) — Participant experienced breathing issues related to sinus infection.
orthopedic (Surgical and medical procedures) | 0 (0) | 1 (1) — wrist pain following surgery

LIMITATIONS AND CAVEATS:
Study sample lacked racial, ethnic and gender diversity. The study was on-going during COVID-19 closures which impacted participants' ability to take part in in-person study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT02719327/Prot_SAP_000.pdf